CLINICAL TRIAL: NCT04792671
Title: Prevalence and Risk Factors of Women Mental Health Disorders in Assiut Governorate
Brief Title: Prevalence and Risk Factors of Women Mental Health Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer, resarcher OF Neurology and Psychiatry department, Assiut University
Other Study IDs: women mental health disorders
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Psychiatric Problem; Wolman Disease
Keywords: women; mental health
MeSH Terms: conditions — Wolman Disease; Psychological Well-Being | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perinatal group: females who are pregnancy
  Interventions: Behavioral: Sociodemographic variables; Behavioral: Family affluence scale (FAS); Behavioral: Edinburgh postnatal depression scale (EPDS); Behavioral: Symptom Checklist 90 "SCL 90":
- postpartum group: female who get delivery(from day 1 up to 1 year)
  Interventions: Behavioral: Sociodemographic variables; Behavioral: Family affluence scale (FAS); Behavioral: Edinburgh postnatal depression scale (EPDS); Behavioral: Symptom Checklist 90 "SCL 90":

INTERVENTIONS:
Behavioral: Sociodemographic variables — age, residence, education of the mother and her husband, occupation of the mother and her husband, parity, gender, and age of the last baby.
Behavioral: Family affluence scale (FAS) — a four-item measure of family wealth, has been developed in the WHO Health Behaviour in School-aged Children Study as an alternative measure.
Behavioral: Edinburgh postnatal depression scale (EPDS) — s a questionnaire originally developed to assist in identifying possible symptoms of depression in the postnatal period. It also has adequate sensitivity and specificity to identify depressive symptoms in the antenatal period and is useful in identifying symptoms of anxiety. more than 9 is clinically diagnosed
Behavioral: Symptom Checklist 90 "SCL 90": — is a 90-item questionnaire used to assess psychological problems. It is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. More than 60 is considered clinically diagnosed

SUMMARY:
Perinatal major depressive disorder affects 20% of women, while perinatal anxiety affects 10% of women. Although pharmacological treatment has shown effectiveness, many pregnant women are concerned about potential adverse effects on the fetus, maternal-infant bonding, and child development.. On the other hand, Depressive disorder in women mainly occurs during the first year after childbirth. It takes many forms according to the onset, severity, and duration of the symptoms including; Postpartum blues (PPB), Postpartum depression (PPD), and Postpartum psychosis (PPP). Lack of access to mental health services during the perinatal period is a significant public health concern that may worse outcome.

So, we aimed to study prevalence of women mental health in Assiut governorate and evaluate possible risk factor for it

ELIGIBILITY:
Inclusion Criteria:

* age 18 years -50 years.
* No previous history of psychiatric, neurological or medical disease

Exclusion Criteria:

* intelligence equation less than 80
* have history of psychiatric, neurological or medical disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: This is study will take part in the Assiut government primary health centres in community
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
measure the prevalence of DSM 5 psychiatric disorders in perinatal and postnatal | through study completion, an average of 1 year
measure of risk factor of DSM 5 psychiatric disorders in perinatal and postnatal | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sambrook Smith M, Lawrence V, Sadler E, Easter A. Barriers to accessing mental health services for women with perinatal mental illness: systematic review and meta-synthesis of qualitative studies in the UK. BMJ Open. 2019 Jan 24;9(1):e024803. doi: 10.1136/bmjopen-2018-024803. PMID 30679296
- [Result] Sheffield KM, Woods-Giscombe CL. Efficacy, Feasibility, and Acceptability of Perinatal Yoga on Women's Mental Health and Well-Being: A Systematic Literature Review. J Holist Nurs. 2016 Mar;34(1):64-79. doi: 10.1177/0898010115577976. Epub 2015 Apr 20. PMID 25896571
- [Result] Sharma V, Burt VK. DSM-V: modifying the postpartum-onset specifier to include hypomania. Arch Womens Ment Health. 2011 Feb;14(1):67-9. doi: 10.1007/s00737-010-0182-2. Epub 2010 Sep 25. PMID 20872155